CLINICAL TRIAL: NCT00497653
Title: Determination if Oral DCI Administration to Women With PCOS Increases Total DCI Content in Urine and Blood...
Brief Title: Oral Administration of DCI to Women With PCOS
Acronym: PCOS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2R01HD35629 P2; 2R01HD035629 (NIH)
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DCI (Experimental)
  Interventions: Drug: DCI
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DCI — D-chiro-inositol 1200mg twicely daily for 6 weeks
  Arms: DCI
Drug: Placebo — Placebo, twice daily for 6 weeks
  Arms: Placebo

SUMMARY:
To determine if oral DCI administration to women with PCOS increases the total DCI content in urine and blood, and, if so, if that change is accompanied by i) an increase in DCI-IPG release in blood (as determined by bioactivity) during an oral glucose challenge and ii) an increase in whole-body insulin sensitivity.

DETAILED DESCRIPTION:
A total of 46 women will be studied. We will study 23 obese and 23 non-obese women. There will be no BMI restriction. Twenty-three women will be randomly assigned to receive DCI (experimental group) and 23 women to receive placebo (control group). The women will be studied during the equivalent of the follicular phase of the cycle, as documented by a serum progesterone concentration of 2 ng/ml.

PCOS will be defined using criteria developed at the 1990 NICHD conference on PCOS3 - i.e., all women will have oligomenorrhea (eight or fewer menstrual periods annually) and hyperandrogenemia (elevated serum total or free testosterone concentration), and secondary causes of hyperandrogenism or ovulatory dysfunction will be excluded (see below: Entrance Criteria). All women will undergo a standard oral glucose tolerance test (OGTT) to screen for diabetes mellitus,16 but impaired glucose tolerance (IGT) will not be an exclusion criteria because of the high prevalence of IGT in this population.8,17-19 We intentionally will not screen the women for the presence of insulin resistance. Women with PCOS who have disorders associated with insulin resistance - such as hypertension21-23 or dyslipidemia21-23 - will not be excluded as long as they have been on a stable dose of medication for 6 months.

ELIGIBILITY:
Inclusion Criteria:-

(1) Non-obese and obese women with PCOS between 18-40 years of age. (2) oligomenorrhea ( 8 menstrual periods annually), (3) biochemical hyperandrogenemia (elevated total or free testosterone), (4) normal thyroid function tests and serum prolactin, and (5) exclusion of 21 -hydroxylase deficiency by a fasting 17 -hydroxyprogesterone <200 ng/dl.41 (6) acceptable health on the basis of interview, medical history, physical examination, and laboratory tests (CBC, SMA20, urinalysis). (7) Signed, witnessed informed consent. (8) Ability to comply with study requirements.

Exclusion Criteria: - (1) Diabetes mellitus by fasting glucose or OGTT, or clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, neoplastic and malignant disease (other than non-melanoma skin cancer). (2) Current use of oral contraceptives, DepoProvera or Norplant.. (3) Documented or suspected recent (within one year) history of drug abuse or alcoholism. (4) Ingestion of any investigational drug within two months prior to study onset.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2001-02; Primary Completion 2007-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine if oral DCI administration to women with PCOS increases the total DCI content in urine and blood. | 43 days

CONTACTS AND LOCATIONS:
Overall Officials: John E. Nestler, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- General Clinical Research Center, Richmond, Virginia, United States